CLINICAL TRIAL: NCT04852705
Title: A Multi-national, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of SARS-CoV-2 Vaccine (Vero Cells), Inactivated for the Prevention of COVID-19 in Healthy Adults Aged 18 Years and Older
Brief Title: A Study to Evaluate the Efficacy, Safety and Immunogenicity of SARS-CoV-2 Vaccine (Vero Cells), Inactivated in Healthy Adults Aged 18 Years and Older (COVID-19)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Kangtai Biological Products Co., LTD (Industry)
Collaborators: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021L001
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- candidate vaccine (Experimental)
  Interventions: Biological: SARS-CoV-2 Vaccine (Vero Cells), Inactivated
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 Vaccine (Vero Cells), Inactivated — 2 doses of SARS-CoV-2 Vaccine (Vero Cells), Inactivated should be administered as an intramuscular injection into the lateral deltoid of the upper arm with a 28-day interval.
  Arms: candidate vaccine
Biological: Placebo — 2 doses of Placebo should be administered as an intramuscular injection into the lateral deltoid of the upper arm with a 28-day interval.
  Arms: Placebo

SUMMARY:
The study will be a multi-national, endpoint-driven, randomized, double-blind, placebo-controlled, adaptive study in which participating adults will be randomized 1:1 to receive 2 doses of either candidate vaccine or placebo on Day 0 and 28. A total of 28,000 healthy adults aged 18 years and older will be enrolled and followed for efficacy, safety, and immunogenicity evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy residents ≥ 18 years at the time of consent, be voluntary and capable of signing the informed consent forms.
* Be able to understand and comply with study requirements/ procedures.
* Participants with negative results of SARS-CoV-2 Realtime-PCR (RT-PCR) detection.
* For females or sex-partners of males at childbearing age: be willing to use birth control for 3 months after the 2nd dose.
* For females of childbearing potential (Pausimenia ≤ 2 years ) must: have a negative urine or blood pregnancy test at screening
* Axillary temperature < 37.3℃/99.1℉ when screening (Subsequent measurements of temperature should be performed at the same site per participant; temperature measured by other methods should be converted to axillary temperature ).

Exclusion Criteria:

* Previous treatments for curing or preventing COVID-19 (including vaccination of various COVID-19 vaccines).
* History of Severe Acute Respiratory Syndrome (SARS), Middle East Respiratory Syndrome (MERS) or other coronavirus infections.
* History of allergy to any components of the candidate vaccine or severe allergic reactions to vaccine or medicine (including, but not limited to, allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, or local allergic necrosis (Arthus reaction)).
* Positive for HIV detection.
* History or family history of convulsion, epilepsy, encephalopathy, and psychosis.
* Active stage of malignancies, malignancies without adequate treatments, malignancies with potential risk for recurrence during the study.
* Severe or uncontrolled cardiovascular, neurological, blood and lymphatic, kidney, liver, respiratory, metabolic and skeletal diseases.
* Congenital or functional absence of spleen, complete or partial removal of spleen in any case.
* Chronic administration (defined as ≥ 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the 1st vaccination (eg. corticosteroids, ≥ 0.5 mg/kg/day prednisone or equivalent; but, inhaled and topical steroids are allowed).
* Planned administration/administration of a vaccine not foreseen by the study protocol less than 7 days before 1st dose of candidate vaccine for inactivated vaccines or 14 days before 1st dose of candidate vaccine for attenuated live vaccines.
* Receipt of blood products and/or immunoglobulins within 3 months prior to enrollment or expected receipt during the study.
* Donate or loss ≥ 450 ml of blood within 1 month prior to enrollment, or expected blood donation during the study.
* Fever: axillary temperature ≥ 37.3℃/99.1℉ within the past 24 hours (Subsequent measurements of temperature should be performed at the same site per participant; temperature measured by other methods should be converted to axillary temperature ).
* Those who participated in other clinical trials 1 month prior to the enrollment or used any investigational or non-registered drug during the study period; Those who are unable to finish follow-up or fail in efficacy assessments.
* Breastfeeding females should not be included.
* Ineligible for the study based on the assessment of investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28000 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Incidence density of symptomatic COVID-19 cases | 14 days after full vaccination
  Incidence density of symptomatic COVID-19 cases occurring from 14 days after full vaccination.

SECONDARY OUTCOMES:
Incidence density of COVID-19 moderate cases and above | 14 days after full vaccination
  Incidence density of COVID-19 moderate cases and above occurring from 14 days after full vaccination.
Incidence density of COVID-19 severe cases and above | 14 days after full vaccination
  Incidence density of COVID-19 severe cases and above occurring from 14 days after full vaccination.
Incidence density of COVID-19 death cases and above | 14 days after full vaccination
  Incidence density of COVID-19 death cases and above occurring from 14 days after full vaccination.
Incidence density of symptomatic COVID-19 cases in different age groups | 14 days after full vaccination
  Incidence density of symptomatic COVID-19 cases occurring from 14 days after full vaccination in different age groups (18~59 years and ≥ 60 years).
Incidence of solicited local adverse events | 0-7 days after each vaccination
  Incidence of solicited local adverse events occurring 0-7 days after each vaccination.
Incidence of solicited general adverse events | 0-7 days after each vaccination
  Incidence of solicited general adverse events occurring 0-7 days after each vaccination.
Incidence of unsolicited adverse events | 0-28 days after each vaccination
  Incidence of unsolicited adverse events occurring 0-28 days after each vaccination.
Incidence of SAE | from the 1st dose through the end of study
  Incidence of SAE occurring from the 1st dose through the end of study.
Incidence of AESI | from the 1st dose through the end of study
  Incidence of AESI occurring from the 1st dose through the end of study.
Seroconversion rate of SARS-CoV-2 neutralizing antibody | 28 days, 90 days, 180 days and 360 days after full vaccination
  Seroconversion rate of SARS-CoV-2 neutralizing antibody in the immunogenicity subgroup
Geometric mean titer of SARS-CoV-2 neutralizing antibody | 28 days, 90 days, 180 days and 360 days after full vaccination
  geometric mean titer of SARS-CoV-2 neutralizing antibody in the immunogenicity subgroup
Geometric mean fold increase of SARS-CoV-2 neutralizing antibody | 28 days, 90 days, 180 days and 360 days after full vaccination
  Geometric mean fold increase of SARS-CoV-2 neutralizing antibody in the immunogenicity subgroup
Seroconversion rate of SARS-CoV-2 IgG binding antibody | 28 days, 90 days, 180 days and 360 days after full vaccination
  Seroconversion rate of SARS-CoV-2 IgG binding antibody in the immunogenicity subgroup
Geometric mean titer of SARS-CoV-2 IgG binding antibody | 28 days, 90 days, 180 days and 360 days after full vaccination
  Geometric mean titer of SARS-CoV-2 IgG binding antibody in the immunogenicity subgroup
Geometric mean fold increase of SARS-CoV-2 IgG binding antibody | 28 days, 90 days, 180 days and 360 days after full vaccination
  Geometric mean fold increase of SARS-CoV-2 IgG binding antibody in the immunogenicity subgroup